CLINICAL TRIAL: NCT02471287
Title: The Genetics of Inherited Eye Disease
Brief Title: Genetics of Inherited Eye Disease
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150128; 15-EI-0128
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09-30

CONDITIONS: Genetic Eye Disease
Keywords: Rare; Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected Participants: Participants with eye disease
- Healthy volunteers: Unaffected first degree relatives of participants with a known or suspected inherited eye disease.

SUMMARY:
Background:

Research has identified some of the genes involved in inherited eye diseases. But for many of these diseases, the genes are not yet known. Researchers want to try to find these genes. They also hope to learn more about how symptoms differ in people with similar gene changes.

Objective:

To learn more about genes involved in eye diseases.

Eligibility:

People who have a known or suspected inherited eye disease, and their relatives.

Design:

* All participants will have a medical history, physical exam, and eye exam. They will have blood taken.
* Participants with an eye disease may have eye cell samples taken using a swab or biopsy procedure.
* Participants may have a skin biopsy. A 3mm piece of skin will be removed.
* Participants may provide samples of tears, urine, saliva, stool, hair, or inner cheek cells.
* Participants may have a retina test. They may also have a test that uses light to measure retina thickness.
* Participants may have an eye movement test. Electrodes will be placed on the skin next to both eyes.
* Participants may have a fluorescein angiography. A dye will be given through an intravenous line in the arm. A camera will take pictures of the dye as it flows through the eyes blood vessels.
* Participants may have microperimetry. They will sit at a computer screen and press a button when they see a light.
* Participants may have an eye movement test. They will wear contact lenses or goggles and watch a series of spots on a computer screen.
* Participants may complete a color vision test.
* Participants will provide a specimen for genetic testing.
* Participants may have a MRI.
* Participants may complete questionnaires.

DETAILED DESCRIPTION:
OBJECTIVE:

Molecular genetics and genomics are revolutionizing the delivery of medicine in general and ophthalmology in particular. New treatment and prevention strategies rely on a detailed understanding of the genetics and molecular pathogenesis of vision-threatening disease. In addition, in order to determine whether an intervention is therapeutic, we must first have some understanding of what the best clinical outcome variables are for measuring a treatment effect. Because our ultimate goal is to develop disease-specific protocols for specific inherited conditions, establishing this protocol will help us establish an initial critical mass of patients and of knowledge to write such protocols; as such, this protocol will be hypothesis generating. A secondary aim of this protocol is to provide a mechanism for obtaining research samples from subjects that may be used for laboratory investigations; in this case, the basic research may be both hypothesis generating and/or hypothesis testing. Lastly, the Ophthalmic Genetics Branch, as a leader in the field and a sponsor of a clinical training program, should have the ability to serve as a tertiary referral center for the nation in the area of undiagnosed genetic eye diseases.

STUDY POPULATION:

One thousand one hundred (1100) individuals with inherited eye diseases and 400 healthy volunteers (the unaffected relatives of affected participants) will be enrolled.

DESIGN:

This is a combined evaluation/treatment protocol and a genetic repository study. In general, participants will undergo a complete, age-appropriate, baseline examination and may provide a blood or saliva sample. Some participants may undergo more specialized ophthalmic and/or systemic testing, if clinically indicated by the investigator. Data and specimens generated through clinical care procedures may be collected and analyzed. The data and images obtained from these tests may be used for determining eligibility into another NEI protocol. Additionally, the collection of these data will help meet the primary research objectives of this study. Participants may be asked to complete optional participant reported outcome (PRO) questionnaires which will be assigned based on current diagnosis and previous testing. In a small number of cases, collection of blood, readily available biospecimens and body fluids (e.g., urine, saliva, tear fluid, stool, hair or cheek swab samples), conjunctival swab or lacrimal gland biopsy, impression cytology, and/or a punch skin biopsy may also be performed for research purposes.

OUTCOME MEASURES:

Given the breadth of ages and disease processes covered under this protocol, we will not systematically obtain any single outcome variable beyond visual acuity on research subjects. However, detailed, disease-specific findings will be collected through the NEI electronic medical record. Findings from systemic testing and from outside exams may be tabulated in a separate, secure database in the laboratory of the Principal Investigator (PI).

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they:

1. Have a known or suspected inherited eye disease OR are an unaffected (usually first degree) relative of a participant with a known or suspected inherited eye disease.
2. Have the ability to cooperate with an age-appropriate eye exam.
3. Have the ability to understand and sign an informed consent or have a parent/legal guardian to do so if they are minor children or have a legally authorized representative if they are adults without consent capacity. Unaffected adult relatives of a participant should be able

to provide consent.

EXCLUSION CRITERIA:

Participants will not be eligible if:

1. They are unwilling or unable to be followed as clinically indicated.
2. They have a clear, non-genetic disease etiology (unless they are an unaffected relative).
3. Their participation would not contribute to the NEI research mission, at the discretion of the PI.

Exclusion Criteria for MRI (if applicable)

Participants will not be eligible for optional MRI procedure if:

1. They have metal in their body which would make having an MRI scan unsafe, such as pacemakers, stimulators, pumps, aneurysm clips, metallic prostheses, artificial heart valves, cochlear implants or shrapnel fragments, or if they were a welder or metal worker, since they may small metal fragments in the eye.
2. They have claustrophobia and would feel uncomfortable in the MRI machine.
3. They are not able to lie comfortably on their back for up to one (1) hour.

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1500 participants may be enrolled into this study. One thousand one-hundred (1,100) participants with known or suspected eye diseases and 400 healthy volunteers (unaffected relatives of affected participants) will be accrued for this study. Self-referral is permitted and participants may enroll as a referral from another NEI study.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-06-22 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Establish cohort | Ongoing
  Establish an initial "critical mass" of participants and knowledge to develop disease-specific protocols for specific inherited eye conditions.

SECONDARY OUTCOMES:
Suggest best clinical outcome measures | ongoing
  Suggesting the best clinical outcome measures to follow patients with various inherited eye diseases
Revealing systematic comorbidities | ongoing
  Revealing systemic comorbidities that occur in patients with various inherited eye diseases.
Provide a mechanism for collecting biological samples | ongoing
  Provide a mechanism for collecting biological samples from well-phenotyped subjects for basic laboratory research
Determine the genetic cause(s) and molecular pathogenesis | ongoing
  Determine the genetic causes(s) and molecular pathogenesis of a known or suspected inherited disorder of vision in an individual patient and his/her family.

CONTACTS AND LOCATIONS:
Overall Officials: Laryssa A Huryn, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bender C, Woo EG, Guan B, Ullah E, Feng E, Turriff A, Tumminia SJ, Sieving PA, Cukras CA, Hufnagel RB. Predominant Founder Effect among Recurrent Pathogenic Variants for an X-Linked Disorder. Genes (Basel). 2022 Apr 12;13(4):675. doi: 10.3390/genes13040675. PMID 35456481
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-EI-0128.html